CLINICAL TRIAL: NCT06106087
Title: Supporting Healthcare Improvement Through Facilitation & Training
Acronym: SHIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Health (Unknown)
Responsible Party: Principal Investigator, Malcolm Doupe, Associate Professor, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H2023:258
Record Dates: First submitted 2023-10-04; First posted 2023-10-30 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Frontline Staff Working Within Personal Care Home Facilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QI Training (Other): Frontline staff in personal care homes will receive quality improvement training from an experienced quality advisor and support staff in making changes aimed to improve the quality of care for residents in the home.
  Interventions: Other: Mixed methods quality improvement intervention

INTERVENTIONS:
Other: Mixed methods quality improvement intervention — Quality improvement training for frontline PCH staff

SUMMARY:
SHIFT will support personal care home (PCH) staff to conduct quality improvement (QI) initiatives more purposefully and objectively in their regular care setting in ways that help to sustainably improve the quality of care and/or life of residents.

DETAILED DESCRIPTION:
The SHIFT study will take place at approximately thirteen (13) residential long-term care facilities in Manitoba during a one-year period. These sites will be licensed by the provincial government and provide 24-hours on-site housing and health care services for older adults by professional (nursing) staff, allied health care professionals and unregulated staff.

In consultation with SHIFT research staff, a senior administrator at each facility will be identified to take on the role of Senior Sponsor (e.g. Director of Care, CEO) for the project. Quality improvement (QI) teams will be formed at each site and team formation will also occur in consultation with research staff. QI teams will have 5-6 participants comprised of a Team Sponsor (e.g. Unit Manager) and Team Members (e.g., Care Aides and Allied Staff).

The SHIFT intervention is comprised of three major components that include:

1. PDSA (plan-do-study-act) Facilitation comprised of workshops interspersed with site-specific (i.e., context-sensitive) coaching sessions designed to help team members plan for and ably conduct their PDSA innovations;
2. Readiness for Change Activities designed to help SHIFT team members more purposefully prepare for the intervention (e.g., by selecting PCH units with the appropriate personnel and context to participate in SHIFT, recruiting team members with the appropriate knowledge and social capital to help ensure project success); and,
3. LeaderShift Modules designed to help Team Sponsors more effectively support front-line team members to plan, implement, and evaluate their SHIFT PDSA cycles.

ELIGIBILITY:
Facility Inclusion Criteria:

* A personal care home (PCH) which provides 24-hour on-site housing and health care services care for older adults by professional (nursing) staff and others.
* Located in Manitoba.
* Licensed by the provincial government.
* 90% of residents aged 65 or over.
* Facility operations conducted in the English language.

Facility Exclusion Criteria:

* Chronic care facilities.
* Transition care facilities.
* Facilities that are expected to undergo major changes during the study intervention (e.g., where a unit is expected to close or the site is expected to undergo major renovations).

Individual Staff Inclusion Criteria:

* have worked on the unit for a minimum of three months.
* have worked at least 6 shifts per month on the unit.
* be able to travel to workshops and participate in relevant SHIFT activities.
* work well with other team members.
* have the respect of staff on the unit.
* be able to communicate effectively with colleagues.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-11-03 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Team fidelity to the quality improvement implementation process | Through study completion, an average of 8 months
  Frontline teams will implement their change ideas using iterative plan-do-study-act (PDSA) cycles. Each team's progress will be captured by the SHIFT quality advisor during regular meetings. After each meeting the quality advisor will complete a structured diary that captures each team's PDSA process using a published scoring system (DOI: org/10.1186/s40814-022-00975-8). This tool measures the appropriateness of each team's aim statement (e.g., being specific, having timeframes), assesses their ability to properly measure and interpret data (e.g., documents pain reduction using run charts) to guide next PDSA steps, and reports the number of PDSA cycles they completed. As described in the aforementioned manuscript, multiple researchers will judge each team's progress independently and then meet to reach consensus opinion.
Level of readiness for change (R4C) among study participants | Baseline
  Each participant will complete a baseline survey to assess their R4C. This survey uses questions from existing tools modified for our target group. It will assess people's perceived R4C at the macro (e.g. "SHIFT aligns with our health system priorities"), meso (e.g. "SHIFT is viewed strongly by leaders at my site"), and micro level (e.g. "I have the skills to conduct SHIFT").
  Team R4C scores will be correlated with results of Outcome Measure 1 (team fidelity to the implementation process) to descriptively assess if teams with higher baseline R4C scores make better PDSA progress.
Identifying readiness for change (R4C) attributes that are precursors to PDSA implementation success. | End of study (after an average of 8 months)
  While readiness for change (R4C) is a well-established concept, it is unclear if and how these processes help teams be more successful. At study start participants will engage in R4C discussions to understand their role in SHIFT, responsibilities and time required, and supports available.
  During focus groups at study end, we will ask participants to (1) reflect on preparatory R4C activities, and (2) compare these to their SHIFT experiences including successes and challenges they encountered. During these focus groups people will suggest additional R4C activities that would have helped them to better prepare for SHIFT.
Value of the LeaderShift program from the perspective of participants | End of study (after an average of 8 months)
  We are developing a novel leadership program (called LeaderShift) that teaches formal nursing home leaders how to help their staff conduct quality improvement initiatives more effectively. LeaderShift training includes four instructional workshops and two 1-1 coaching sessions throughout the study to help participants apply lessons during daily routines. Participants will discuss the value of LeaderShift with researchers in an end-of-project focus group to examine its value, to discuss components that were more and less effective, and to make suggestions for improving LeaderShift content. Following the principles employed by others (doi.org/10.1016/j.jcjq.2018.04.009) focus group data will be analyzed using qualitative constant comparative analysis to understand the extent, properties, and processes related to LeaderShift program success.
Participant Fidelity to the LeaderShift Program | Through study completion, average of 8 months
  LeaderShift is based on the LEADS framework that coaches people to lead in complex systems (DOI: 10.1108/LHS-02-2017-0002) and instructs people how to (1) develop key leadership characteristics (the domain of "Leading Self" in LEADS), (2) help others achieve their goals ("Engage Others"), and (3) create an environment of continuous improvement ("Systems Transformation"). Coaching will be provided during workshops and 1:1 sessions to discuss leadership change progress and to provide additional training where needed. After each session the LeaderShift coach will complete a semi structured diary documenting each participant's progress made with implementing these leadership principles. This will include a Likert Scale score of 0 (no success) to 9 (complete success) indicating the extent of participant progress and an explanation of the score provided. Researchers will review the diaries for each participant independently and develop a consensus score demonstrating overall success.
Changes in leadership approaches witnessed by frontline teams | End of study (after an average of 8 months)
  During end-of-study focus groups we will ask frontline team members if they noticed changes in their Team Sponsor's (direct supervisor's) leadership approach, to provide examples explaining these changes, and to discuss if and how this helped them to achieve PDSA success. Data will be presented aggregately across all SHIFT teams combined.

SECONDARY OUTCOMES:
Improvement in resident care perceived by team members. | End of study (after an average of 8 months)
  Each team will participate in an end-of-study focus group where members will be asked to reflect on their change ideas and discuss how these ideas improved resident care. Teams will be asked to provide examples illustrating how residents benefited from their change ideas. Following the principles employed by others (doi.org/10.1016/j.jcjq.2018.04.009) focus group data will be analyzed using a qualitative constant comparative analysis technique to understand the properties, processes, and causes of each team's perceived success.

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Doupe, Phd, Principal Investigator — University of Manitoba
Locations (1):
- Winnipeg Regional Health Authority, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No